CLINICAL TRIAL: NCT06008119
Title: A Multicenter, Randomized, Open-label, Phase 3 Study to Evaluate the Efficacy and Safety of Tunlametinib Plus Vemurafenib in Patients With BRAF V600E-mutant Metastatic Colorectal Cancer
Brief Title: Efficacy and Safety of Tunlametinib Plus Vemurafenib in Patients With BRAF V600E-mutant Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-304
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer Metastatic
Keywords: BRAFV600E mutant
MeSH Terms: interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Tunlamatinib plus Vemurafenib
  Interventions: Drug: Tunlametinib plus Vemurafenib
- Control (Active Comparator): Investigators' choice
  Interventions: Drug: Doublets Chemotherapy ± Bevacizumab or Doublets Chemotherapy ± Cetuximab

INTERVENTIONS:
Drug: Tunlametinib plus Vemurafenib — 12mg BID Tunlametinib+720mg BID Vemurafenib
  Arms: Experimental
Drug: Doublets Chemotherapy ± Bevacizumab or Doublets Chemotherapy ± Cetuximab — According to investigators' suggestion
  Arms: Control

SUMMARY:
This is a multicenter, randomized, open-label, Phase 3 study

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, Phase 3 study to evaluate Tunlamatinib plus Vemurafenib versus Investigator's choice of Chemotherapy based treatment as controls in patients with BRAFV600E mutant Metastatic Colorectal Cancer (CRC) whose disease has progressed after 1 or more prior regimens in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Before study entry, written informed consent must be obtained from the patient prior to performing any study-related procedures.
  2. Male or female patients with 18 to 70 years of age at time of informed consent;
  3. Histological or cytologically confirmed metastatic CRC
  4. Presence of BRAFV600E in tumor tissue as previously determined by a local assay at any time prior to Screening or by the central laboratory (BRAFV600 is permitted)
  5. Able to provide a sufficient amount of representative tumor specimen (primary or metastatic, archival or newly obtained) for confirmatory central laboratory testing of BRAF mutation status.
  6. Progression of disease after 1 or more prior regimens in the metastatic setting
  7. At least 1 site of radiographically measurable disease by RECIST 1.1
  8. Eastern Cooperative Oncology Group (ECOG) Performance Status(PS) of 0 to 1;
  9. Life expectancy ≥ 3 months;
  10. Can swallow the medicine,
  11. Adequate hematologic, renal, cardiac and liver function as defined by laboratory values performed within 7 days prior to initiation of dosing:
  12. Be willing and able to complete all the study procedures and follow-up examinations.

Exclusion Criteria:

* Exclusion Criteria:

  1. Prior treatment with any BRAF and MEK inhibitor;
  2. Known contraindication to receive the treatment of control arm (according to latest PI).
  3. Symptomatic brain metastasis or leptomeningeal disease
  4. History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to randomization
  5. Known history of acute or chronic pancreatitis
  6. Uncontrolled GI bleeding, Dysphagia，refractory nausea, vomiting, small bowel resection or any other gastrointestinal ailment that would preclude study drug absorption.
  7. Serious cardiovascular disease , including uncontrolled congestive heart failure, uncontrolled hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia , deep vein thrombosis or pulmonary emboli or cerebrovascular events ≤ 6 months prior to starting study treatment;
  8. History or current evidence of retinal vein occlusion or current risk factors for retinal vein occlusion (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
  9. Concurrent neuromuscular disorder that is associated with the potential of elevated creatine (phosphor)kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
  10. Uncontrolled blood pressure despite medical treatment
  11. Concurrent or previous other malignancy within 5 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy
  12. Residual common terminology criteria for adverse events (CTCAE) ≥ Grade 2 toxicity from any prior anticancer therapy, with the exception of Grade 2 alopecia or Grade 2 neuropathy
  13. Anti-HIV(+) , Anti-TP( +); Active hepatitis B or hepatitis C infection …….

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 12 months
  defined as the time from first dose to the earliest documented disease progression or death due to any cause

SECONDARY OUTCOMES:
Overall Survival（OS） | up to 12 months
  defined as the time from the date of taking drugs to the date of death due to any cause
Overall Response Rate（ORR） | up to 12 months
  Defined as the proportion of subjects with an optimal response of CR or PR over the course of the study from enrollment to disease progression
Duration of Response（DOR） | up to 12 months
  Defined as the time from the first CR or PR evaluation of tumor efficacy to the first occurrence of PD or death from any cause (whichever occurs first)
Disease control rate (DCR) | up to 12 months
  roportion of subjects with response defined as CR, PR, and SD throughout the study from subjects first dose to disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Oncology Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No